CLINICAL TRIAL: NCT01787396
Title: A Multicenter, Randomized, Active-controlled, Parallel Group, Double-blind, Phase III Trial to Evaluate the Efficacy and Safety of Initial Combination Therapy With Gemigliptin 50mg q.d and Metformin q.d Compared With Either Monotherapy in Treatment naïve Patients With Type 2 Diabetes
Brief Title: Phase III Trial to Evaluate the Efficacy and Safety of Initial Combination Therapy With Gemigliptin 50mg q.d and Metformin q.d
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LG-DPCL011
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LC15-0444; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Arm1 (Experimental): Gemigliptin 50mg + Metformin Once daily with dinner
  Interventions: Drug: Gemigliptin 50mg; Drug: Metformin
- Arm 2 (Experimental): Gemigliptin 50mg + Placebo(Metformin)Once daily with dinner
  Interventions: Drug: Gemigliptin 50mg; Drug: Placebo(Metformin)
- Arm3 (Experimental): Metformin+ Placebo(Gemigliptin 50mg)Once daily with dinner
  Interventions: Drug: Metformin; Drug: Placebo(Gemigliptin)

INTERVENTIONS:
Drug: Gemigliptin 50mg
  Arms: Arm 2; Arm1
Drug: Placebo(Metformin)
  Arms: Arm 2
Drug: Metformin
  Arms: Arm1; Arm3
Drug: Placebo(Gemigliptin)
  Arms: Arm3

SUMMARY:
The objective of this study is to evaluate efficacy and safety of initial combination therapy with Gemigliptin 50mg q.d and Metformin q.d compared with either monotherapy in treatment naïve patients with type 2 diabetes, In other words, to proof superiority of initial combination therapy with Gemigliptin and Metformin than each monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 2 diabetes mellitus
2. Adults over 20 of age
3. Patients with hemoglobin A1c (HbA1c) over 7.5% at Visit1(screening) and no previous antidiabetic drugs before Visit 1(screening) or patients with hemoglobin A1c (HbA1c) between 7%~10.5%, Patients treated with metformin monotherapy before Visit 1(screening).

   Patients with no previous antidiabetic drugs
4. Patients with hemoglobin A1c (HbA1c) between 7.5%~11% at Visit 2(randomization)

Exclusion Criteria:

1. Patients with type 1 diabetes mellitus Diabetic ketoacidosis or Hyperosmolar non-ketotic coma.
2. Patients with gestational diabetes, or secondary diabetes
3. Patients with New York Heart Association (NYHA) class III-IV congestive heart failure or patients with arrhythmia requiring treatment
4. Patients with dysfunctional thyroid gland (with abnormal level of TSH)
5. Patients with active bladder cancer.
6. Tests which need to be given radiation iodide dye by intravenous.(ex, intravenous urography, intravenous cholangiography, angiography, CT with dye)
7. Severe infection, pre or post operation.(Simple surgery which does not have restriction of food and fluid), severe trauma patient.
8. Patients with pituitary insufficiency or adrenal dysfunction.
9. Patients with pulmonary infarction, severe pulmonary dysfunction, hypoxemia.
10. Patients with gastrointestinal disorders(ex. Dehydration, Diarrhea, Vomiting)
11. Female patients who is gravida or in lactiferous phase or confirmed pregnancy by serum or urine.
12. Patients with body mass index (BMI) below 20 kg/m2 or exceeding 40 kg/m2
13. Male patients with Serum Creatinine level over 1.5mg/dl, Female patients with serum creatinine over 1.4mg/dl.
14. Patients with alanine aminotransferase (ALT), aspartate aminotransferase (AST), exceeding 2.5 times or bilirubin exceeding 1.5 times of the upper limit of the normal range
15. Patients who were taking or needed to take any drugs that may affect the control of blood glucose significantly (ex. glucocorticoids)
16. Patients taking thyroid hormone, warfarin, dicoumarin or digoxin.
17. Patients taking CYP3A4 inducers.(ex, Rifampicin(Rifampin), Dexametha-sone, Phenytoin, Carbamazepine, Rifabutin, Phenobarbital)
18. Patients taking Furocemide, Nifedipine, Cimetidine
19. Patients who were treated with Anti-obesity drugs in the last 12 weeks prior to Visit 1(screening)
20. Patients who were treated with insulin or glucagon-like peptide-1 (GLP-1) analogue or in the last 6 months prior to Visit 1.
21. Patients who had experienced myocardial infarction, unstable angina or prior history of coronary artery bypass surgery within 6 months prior to Visit1(screening), or patients with arrhythmia requiring treatment
22. Patients with history of addiction to alcohol or drugs within 1year prior to Visit 1(screening).
23. Patients with history of Diabetic ketoacidosis or Hyperosmolar non-ketotic coma.
24. Patients with history of hypersensitivity to gemiglpitin or Dipeptidyl-peptidase4(DPP4) inhibitors.
25. Patients with history of hypersensitivity to metformin or biguanides.
26. Patients with history of hypersensitivity to Pioglitazone HCl or Thiazolidinediones
27. Patients who participated in other clinical trial within 3 months prior to Visit1(screening).
28. Patients with other reasons who the investigator decided not to be eligible for the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
HbA1c | 24weeks
  Evaluation variables at week 24 to baseline(Visit 2(randomization), week 0)

CONTACTS AND LOCATIONS:
Locations (1):
- LG Life Sciences, Seoul, South Korea